CLINICAL TRIAL: NCT06611683
Title: Effect of Inspiratory Muscle Training on Ventilated Patients in an Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Zuoying Armed Forces General Hospital (Unknown); Kaohsiung Chang Gung Memorial Hospital,Taiwan (Unknown)
Responsible Party: Principal Investigator, Hui-Ling Lin, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAFGHIRB107-027
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Critically Ill, Subacute Adult Patients; Mechanically Ventilation
Keywords: sub-acute critical ill; mechanical ventilation; respiratory muscle training; respiratory muscle strength; rapid shallow breathing index
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inspiratory Muscle Training (Experimental): Subjects received inspiratory muscle training twice daily over five consecutive days, followed by a two-day rest period. This regimen was continued for three consecutive weeks or until the subject no longer required ventilator support.
  Interventions: Procedure: Inspiratory muscle training
- Non-inspiratory muscle training (Sham Comparator): Subjects received routine care.
  Interventions: Procedure: Routine care

INTERVENTIONS:
Procedure: Inspiratory muscle training — A threshold inspiratory muscule device used a starting resistance set at 30% maximum inspiratory pressure, connecting to subject artificial airway. The subjects were then instructed to perform fast and forceful inspirations against added inspiratory resistance. The inspiratory muscle training was conducted twice daily over five consecutive days, followed by a two-day rest period. This regimen continued for three consecutive weeks or until the subject no longer required ventilator support.
  Arms: Inspiratory Muscle Training
Procedure: Routine care — Subjects received routine care without intervention.
  Arms: Non-inspiratory muscle training

SUMMARY:
The goal of this clinical trial is to learn if inspiratory muscle training facilite the liberation of mechanical ventilation. The main questions it aims to answer are:

Does inspiratory muscle training facilitate weaning from mechanical ventilation and enhance muscle strength in critically ill, subacute adult patients?

The main questions it aims to answer are:

Does pulmonary rehabilitation facilitate wwaning form mechanical patients? Does the intervention improve respiratory muscle strength and respiratory patterns?

Participants received:

Inspriatory muscle training twice daily for three consecutive weeks or until the subject no longer required ventilator support.

DETAILED DESCRIPTION:
Patients on mechanical ventilation often experience rapid diaphragm atrophy on the second day, resulting in muscle fiber changes, respiratory muscle weakness. Clinical studies have explored enhancing diaphragm and respiratory muscle strength and endurance through inspiratory muscle, expiratory muscle, and combined respiratory muscle training. This study was to determine if inspiratory muscle training significantly facilitates liberation from mechanical ventilation and improves muscle strength when compared to without IMT among subacute critically ill adult patients.

ELIGIBILITY:
Inclusion Criteria:

* requiring invasive mechanical ventilation for 2 days in an ICU

Exclusion Criteria:

* hemodynamic instability (heart rate 120 beats/min, unstable blood pressure, vasopressor infusion)
* inadequate oxygenation (PEEP 8 cmH2O, FiO2 50%)
* body temperature 38.5°C
* sepsis
* use of sedative infusion
* steroid administration
* home ventilator use before ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of days until liberation from mechanical ventilation | Three weeks
  A record of the number of days until liberation from mechanical ventilation.

SECONDARY OUTCOMES:
Maximum inspiratory pressure | Three weeks
  Maximum inspiratory pressure was measured by having each subject exert maximum inspiratory force against a pressure gauge.
Maximum expiratory pressure | Three weeks
  Maximum expiratory pressure was measured by having each subject exert maximum expiratory force against a pressure gauge.
Peak expiratory flow | Three weeks
  The peak expiratory flow was measured using a respiratory mechanics monitor during three forceful expirations.
Peak inspiratory flow | Three weeks
  The peak inspiratory flow was measured using a respiratory mechanics monitor during three forceful expirations.
Rapid Shallow breathing index | Three weeks
  The RSBI was calculated by dividing the respiratory rate by the tidal volume

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Jane Wang, MS, Study Director — Zuoying Armed Forces General Hospital
Locations (1):
- Zuoying Armed Forces General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The data is available upon request from the principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available 3 three years after the registration
Access Criteria: The data is available upon request from the principal investigator.

REFERENCES:
- [Derived] Wang SJ, Fang TP, Rowley DD, Liu NW, Chen JO, Liu JF, Lin HL. Inspiratory muscle training facilitates liberation from mechanical ventilation in subacute critically ill patients-a randomized controlled trial. Front Med (Lausanne). 2025 Jan 29;11:1503678. doi: 10.3389/fmed.2024.1503678. eCollection 2024. PMID 39944819